CLINICAL TRIAL: NCT07025603
Title: Pilot Evaluation of the Social ABCs Parent-Mediated Intervention for Autistic Toddlers in Israel
Brief Title: Evaluation of the Social ABCs in Israel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Soroka University Medical Center (Other); Azrieli National Centre for Autism and Neurodevelopment Disorders (Unknown)
Responsible Party: Principal Investigator, Judah Koller, Assistant Professor, Clinical Child Psychology and Special Education, Hebrew University of Jerusalem
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020Y1907; SOR-20-0363 (Other: Soroka University Medical Center)
Record Dates: First submitted 2025-06-05; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Autism; Autism Spectrum Disorder (ASD)
Keywords: Social ABCs; Parent-mediated; intervention; Naturalistic Developmental Behavioral Intervention; Pivotal Response Treatment; Early Intervention; Group Intervention; Social Communication
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social ABCs Program Participants (Experimental): All participants will receive the Social ABCs program, a 6-week parent-mediated intervention. Each week includes one group session delivered via Zoom and one to two individual face-to-face coaching sessions with the parent and child. The program teaches parents strategies to support their child's social communication during everyday routines such as play, meals, and caregiving activities.
  Interventions: Behavioral: The social ABCs

INTERVENTIONS:
Behavioral: The social ABCs — The Social ABCs, a parent-mediated intervention for toddlers with suspected or confirmed Autism Spectrum Disorder (ASD), originally developed in Canada (Brian et al., 2016). It is based on principles of Pivotal Response Treatment (PRT, grounded in Applied Behavioural Analysis). The two main goals of the intervention: early functional verbal communication and positive affect sharing in the context of play and caregiving activities.
  The current study follows the Group Social ABCs protocol, a 6-week parent-mediated intervention designed to support early social communication in young children with autism. The program is delivered at two research sites: Soroka and Hebrew University of Jerusalem. Each week, parents participate in: One group session via Zoom, led by a trained Social ABCs coach, with 3-5 parents per group. These sessions introduce strategies and provide peer support, and one to two individual face-to-face coach (See #17-745 for more information).

SUMMARY:
The goal of this study is to evaluate the effectiveness of the Social ABCs program for young autistic children and their parents. The study will also explore predictors of treatment success and child outcomes.

The main questions it aims to answer are:

* Does the Social ABCs program help children use more words and communicate better?
* Does the program help parents feel more confident and less stressed?
* Which children and parents benefit most from the program?

Participants will:

* Join a 6-week Social ABCs program with weekly group and individual coaching sessions
* Complete assessments before and after the program to see how their child and family are doing
* Take part in short video-recorded play sessions to see how communication changes over time

ELIGIBILITY:
Inclusion Criteria:

* children who met diagnostic criteria for autism according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-V), established by independent gold-standard assessments by both a psychologist and a physician (i.e., child psychiatrist, developmental pediatrician, or child neurologist)
* diagnosis received before 30 months of age.
* full-term birth (36-42 weeks gestation) with birth weight >2500 grams

Exclusion Criteria:

* identifiable neurological, genetic, or severe sensory/motor conditions
* attending a special education kindergarten
* participating in a concurrent parent-mediated intervention.

Ages: 12 Months to 40 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability of the Social ABCs Protocol | immediately after the intervention
  Feasibility will be assessed by tracking recruitment rates, retention throughout the 6-week program, and attendance at both group and individual coaching sessions. Acceptability will be evaluated through parent-reported satisfaction surveys completed at the end of the program, as well as qualitative feedback on the format, content, and delivery of the intervention.
The Hebrew Communicative Development Inventory (HCDI). | Baseline (pre-intervention); 6 weeks post-intervention
  The HCDI is the adapted Hebrew version of the MacArthur Communicative Development Inventory (MCDI). The MCDI is a well normed, reliable, and valid tool for vocabulary assessment (Bates et al., 1994). The HCDI is a reliable and sensitive measure of lexical development and emergent grammar, capturing wide variability among Israeli toddlers (Maital et al., 2000). We utilized two versions of the inventory: Words & Gestures for toddlers up to 25 months and Words & Sentences for children 25 months and older. This questionnaire relies on caregiver report to assess children's receptive and expressive vocabulary, speech comprehension, gesture use, morpheme acquisition, and syntactic complexity. In our study, we focused on two variables: receptive vocabulary total score and expressive vocabulary total score
Parenting Stress Index Short Form (PSI-SR). | Baseline (pre-intervention); 6 weeks post-intervention
  The PSI-SR is a self-report, 36-item index of parenting-related stress. Each item is scored on a 5-point Likert-type scale, with higher scores indicating greater parenting stress (range 36-180). Alongside a total stress score, the three subscale scores are derived, each composed of 12 items (range 12-60): parental distress (PD), measuring distress caused by the burdens and restrictions of childcare and personal stressors (e.g., depression, conflict with partner); parent-child dysfunctional interaction (PCDI), assessing parents' negative perception of their interactions with the child and the degree to which the child does not meet their expectations; and difficult child (DC), measuring parents' views of the child's self-regulatory functioning. It also includes a defensive responding scale (DR; seven items, range 7-35), which assesses if the parent is trying to deny or minimize problems.

SECONDARY OUTCOMES:
Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2; Lord et al., 2012). | Baseline (pre-intervention); 6 weeks post-intervention
  This is a semi-structured, standardized behavioral assessment of social communication abilities and restricted and repetitive behaviors. We used the ADOS-2 calibrated severity scores (CSS) to estimate autism symptom severity while separating CSS into the Social Affect (SA) and the Restricted and Repetitive Behavior (RRB) domains. The CSS were specifically developed to enable comparison of autism severity independent of the child's age and language abilities (Hus et al., 2014).
  Verbal ability was evaluated using item A1 of the ADOS-2
The Mullen Scales of Early Learning (MSEL; Mullen, 1995). | Baseline (pre-intervention); 6 weeks post-intervention
  The MSEL is a standardized developmental assessment that quantifies expressive and receptive language, motor, perceptual abilities, and motor development. All MSEL were administered and/or supervised by licensed developmental psychologists.
Adaptive Behavior Assessment System-Second Edition Parent Form, Ages 0-5 (ABAS-II; Harrison & Oakland, 2000). | Baseline (pre-intervention); 6 weeks post-intervention
  The ABAS-II Parent Form (ages 0-5) is a comprehensive norm-referenced parent-report rating scale used for measuring adaptive behaviors and skills in children on a 4-point Likert-type scale, with higher scores indicating better adaptive functioning. The ten skills of the ABAS-II are combined into a general adaptive behavior composite score (GAC) and three composites: conceptual (communication, functional pre-academics, and self-direction), social (social skills and leisure), and practical (self-care, home living, community use, health and safety).
Aberrant Behavior Checklist (ABC; Aman et al., 1985; Kaat et al., 2014). | Baseline (pre-intervention); 6 weeks post-intervention
  The ABC is a caregiver-report measure of disruptive behaviors with 58 items, each rated on a four-point Likert-type scale (0-3), with higher scores indicative of more severe problematic behavior, on five subscales: Irritability (tantrums, aggression and self-injury, 15 items); Social Withdrawal (16 items); Stereotypic Behavior (7 items); Hyperactivity/Noncompliance (16 items); and Inappropriate Speech (4 items). In autistic children, the ABC subscales demonstrate adequate convergent validity (Kaat et al., 2014), however the scale does not have Israeli norms.
Communication and Symbolic Behavior Scales Developmental Profile (CSBS-DP) Infant-Toddler Checklist | Baseline (pre-intervention); 6 weeks post-intervention
  The CSBS-DP Infant-Toddler Checklist is a screening tool designed to determine whether a full developmental evaluation is warranted. It is a parent-report measure, consisting of 24 items that range from a possible of two to four points within each of seven clusters. Scores are given for three composites: Social Composite (Emotion, Eye Gaze, Communication and Gestures Clusters); Speech Composite (Sounds and Words Clusters); Symbolic Composite (Understanding and Object Use Clusters). Norms of the CSBS-DP are available only up to 24 months, so we used the raw scores
Social ABCs Satisfaction Questionnaire (Brian et al., 2016). | immediately after the intervention
  This is a 7-item questionnaire where parents reported whether the intervention was "helpful" in different domains. Ratings were completed using a 5-point scale (1: "not at all helpful" to 5: "extremely helpful").

CONTACTS AND LOCATIONS:
Overall Officials: Judah Koller, PhD, Principal Investigator — Hebrew University of Jerusalem
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Hebrew University of Jerusalem, Jerusalem

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Group Social ABCs Protocol on NIH website — https://clinicaltrials.gov/study/NCT03499262

DOCUMENTS (4):
  • Study Protocol: HUJI (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT07025603/Prot_000.pdf
  • Study Protocol: Soroka (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT07025603/Prot_001.pdf
  • Informed Consent Form: HUJI (2020-07-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT07025603/ICF_002.pdf
  • Informed Consent Form: Soroka (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT07025603/ICF_003.pdf